CLINICAL TRIAL: NCT02003118
Title: A Placebo Controlled, Double Blind, Randomised, 8-week Phase IIa Proof of Concept Study to Assess the Efficacy and Safety of AKR 202 in Patients With Osteoarthritis Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akron Molecules AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AKT-001
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- AKR 202 (Experimental)
  Interventions: Drug: AKR 202
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AKR 202
  Arms: AKR 202
Drug: Placebo
  Arms: Placebo

SUMMARY:
This proof of concept study will be a placebo controlled, randomised, double blind, parallel study. The purpose of the study is to determine efficacy for AKR 202 in the treatment of osteoarthritis (OA) pain in the knee.

ELIGIBILITY:
Inclusion Criteria:

Patient is between 40 and 75 years of age with a clinical diagnosis of OA of the knee for more than 6 months prior to Visit 1 based on clinical and radiographic criteria, and being of American Rheumatism Association (ARA) functional Class I, II, or III. Patients should have an average pain level of between 4 and 8 on a Numeric Rating Scale (NRS) for at least 5 of 7 days before the randomisation, when answering the question: Please, rate the average pain in your index knee during the last 24 hours. Prior to the study, patients should have been using pharmacological treatments, such as Non-Steroidal Anti-Inflammatory Drug (NSAIDs), acetaminophen or weak opioids for their OA pain on a regular basis (defined as having used NSAIDs, acetaminophen or weak opioids at least 10 days out of 30 days during the last month prior to the screening visit).

Exclusion Criteria:

Patient has a concurrent medical/arthritic disease that could confound or interfere with evaluation of efficacy.

Patients with impaired renal function, defined as an estimated creatinine clearance less than or equal to 50 ml/min, or patients taking medications that might impair renal function.

Patient has New York Heart Association (NYHA) Class III-IV congestive heart failure.

The patient has a history of uncontrolled hypertension or a current blood pressure that in the opinion of the Investigator makes the patient unsuitable for the study.

Patients with a trauma or surgery at the index knee within 3 months prior to screening.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
WOMAC | 8 weeks
  Change from baseline in WOMAC pain subscale at Week 8 or at the final visit at the time of patient discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, MD, Study Director — Akron Molecules
Locations (1):
- Clinical study center, Vienna, Austria